CLINICAL TRIAL: NCT04242082
Title: Role of Glucose Transporter (GLUT) Genes Expression in Patients With Psoriasis
Brief Title: Glucose Trnsporter and PEDF in Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SSElkady, Demonstrator at Medical Biochemistry department, Assiut University
Other Study IDs: PGLUTPEDF
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Psoriasis Vulgaris
Keywords: GLUT 1; PEDF; Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will taken from three groups.Then RNA will be extracted,then used for cDNA formation followed by real time PCR to see fold changes of GLUT1 genes expression.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with psoriasis vulgaris only
  Interventions: Diagnostic Test: GLUT 1 gene expression
- patients with psoriasis vulgaris and type 2 diabetes mellitus
  Interventions: Diagnostic Test: GLUT 1 gene expression
- healthy control
  Interventions: Diagnostic Test: GLUT 1 gene expression

INTERVENTIONS:
Diagnostic Test: GLUT 1 gene expression — GLUT 1 gene expression will done on blood samples taken from three groups using real time PCR.
  Pigment epithelium derived factor will used on keratinocytes cell line and compare GLUT 1 gene expression before and after treatment.

SUMMARY:
Psoriasis is a chronic relapsing cutaneous immune mediated inflammatory disease(IMID). In which there are skin lesions characterized by erythema, thickness and scale formation with different size from a pinhead to 20 cm in diameter. Prevalence of psoriasis is 2% to 4% worldwide. Psoriasis occurs at any age with two peaks: between 15-20 years and between 55-60 years. Women are presented with psoriasis at younger age than men ,but with less severity. lesions usually present on knee, elbow, scalp and sacral region this may be attributed to higher traumatic incident .

Psoriasis vulgaris is the most common type, and accounts 90% of cases. Patients with psoriasis vulgaris present with pain, itching and bleeding from skin lesions.

There are many theories for psoriasis pathogenesis: angiogenesis, decrease in apoptosis of keratinocyte, hyperproliferation , alteration of cell to cell adhesion and immune-mediated inflammation.

Patients with immune mediated inflammatory disease (IMID) are susceptible to develop diabetes mellitus, metabolic syndrome, hyperlipidemia, and hypertension.A previous study found that psoriatic patients are more susceptible to type 2 diabetes compared to control.

Glucose transporter type 1(GLUT1) is upregulated in psoriatic patient attributed to angiogenesis and execessive cell proliferation in those patients .Also expression of GLUT 1 is found high with hyperglycemia . A study reported that GLUT 1 density in placenta of women with gestational diabetes was found to be two folds higher than control.

Pigment epithelium derived factor (PEDF) has antiangiogenic effect. Topical application of PEDF on mouse model of psoriatic disease helps in reduction of skin proliferation and angiogenesis.

GLUT 1 overexpression was found to be associated with decrease in PEDF expression in diabetic retinopathy.

In view of that we will compare the level of GLUT 1 gene in psoriatic patients and psoriatic patients with diabetes, as well as healthy control, and detect the effect of PEDF on GLUT 1 expression in vitro using human keratinocytes cell line .

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis vulgaris Patients with psoriasis vulgaris and type 2 diabetes

Exclusion Criteria:

* Factors affect GLUT 1 expression As: tumors either benign or malignant cause increase GLUT 1 expression

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: first group (N=25) : Patients with psoriasis vulgaris second group(N=25) :Patients with psoriasis vulgaris and type 2 diabetes third group(N=25) : healthy control
  data collection :
  * Sex
  * Age
  * BMI
  * Blood glucose level ,HA1c using high performance liquid chromatography (HPLC)
  * Duration of disease (T2D and psoriasis)
  * Severity of psoriasis by psoriasis area severity index (PASI)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-07-31 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
GLUT1 expression in psoriatic patients with or without type 2 diabetes. | through study completion, an average of 2 year
  assessing fold changes of GLUT1 expression in blood samples using real time PCR.
GLUT1 expression in keratinocyte before and after treatment with pigment epithelium derived factor (PEDF) | through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa K Idriss, asst. prof, Study Director — Assiut University; Ayaat ِA Sayed, asst. prof, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abdou AG, Maraee AH, Eltahmoudy M, El-Aziz RA. Immunohistochemical expression of GLUT-1 and Ki-67 in chronic plaque psoriasis. Am J Dermatopathol. 2013 Oct;35(7):731-7. doi: 10.1097/DAD.0b013e3182819da6. PMID 23392136
- [Result] Sondermann W, Djeudeu Deudjui DA, Korber A, Slomiany U, Brinker TJ, Erbel R, Moebus S. Psoriasis, cardiovascular risk factors and metabolic disorders: sex-specific findings of a population-based study. J Eur Acad Dermatol Venereol. 2020 Apr;34(4):779-786. doi: 10.1111/jdv.16029. Epub 2019 Dec 3. PMID 31797464
- [Result] Sarac G, Koca TT, Baglan T. A brief summary of clinical types of psoriasis. North Clin Istanb. 2016 Jun 14;3(1):79-82. doi: 10.14744/nci.2016.16023. eCollection 2016. PMID 28058392
- [Result] Holm JG, Thomsen SF. Type 2 diabetes and psoriasis: links and risks. Psoriasis (Auckl). 2019 Jan 17;9:1-6. doi: 10.2147/PTT.S159163. eCollection 2019. PMID 30697518
- [Result] Granata M, Skarmoutsou E, Trovato C, Rossi GA, Mazzarino MC, D'Amico F. Obesity, Type 1 Diabetes, and Psoriasis: An Autoimmune Triple Flip. Pathobiology. 2017;84(2):71-79. doi: 10.1159/000447777. Epub 2016 Sep 17. PMID 27639922
- [Result] Hagg D, Sundstrom A, Eriksson M, Schmitt-Egenolf M. Severity of Psoriasis Differs Between Men and Women: A Study of the Clinical Outcome Measure Psoriasis Area and Severity Index (PASI) in 5438 Swedish Register Patients. Am J Clin Dermatol. 2017 Aug;18(4):583-590. doi: 10.1007/s40257-017-0274-0. PMID 28342016
- [Result] Li Y, Song Y, Zhu L, Wang X, Yang B, Lu P, Chen Q, Bin L, Deng L. Interferon Kappa Is Up-Regulated in Psoriasis and It Up-Regulates Psoriasis-Associated Cytokines in vivo. Clin Cosmet Investig Dermatol. 2019 Nov 29;12:865-873. doi: 10.2147/CCID.S218243. eCollection 2019. PMID 31819584
- [Result] Matsuura T, Sato M, Nagai K, Sato T, Arito M, Omoteyama K, Suematsu N, Okamoto K, Kato T, Soma Y, Kurokawa MS. Serum peptides as putative modulators of inflammation in psoriasis. J Dermatol Sci. 2017 Jul;87(1):36-49. doi: 10.1016/j.jdermsci.2017.03.014. Epub 2017 Mar 27. PMID 28431948
- [Result] Lee JH, Kim JS, Park SY, Lee YJ. Resveratrol induces human keratinocyte damage via the activation of class III histone deacetylase, Sirt1. Oncol Rep. 2016 Jan;35(1):524-9. doi: 10.3892/or.2015.4332. Epub 2015 Oct 16. PMID 26499368
- [Result] Shaker O, Abdel-Halim M. Connexin 26 in psoriatic skin before and after two conventional therapeutic modalities: methotrexate and PUVA. Eur J Dermatol. 2012 Mar-Apr;22(2):218-24. doi: 10.1684/ejd.2012.1649. PMID 22361809
- [Result] Gaither K, Quraishi AN, Illsley NP. Diabetes alters the expression and activity of the human placental GLUT1 glucose transporter. J Clin Endocrinol Metab. 1999 Feb;84(2):695-701. doi: 10.1210/jcem.84.2.5438. PMID 10022440
- [Result] Calado SM, Alves LS, Simao S, Silva GA. GLUT1 activity contributes to the impairment of PEDF secretion by the RPE. Mol Vis. 2016 Jul 14;22:761-70. eCollection 2016. PMID 27440994
- [Result] Abe R, Yamagishi S, Fujita Y, Hoshina D, Sasaki M, Nakamura K, Matsui T, Shimizu T, Bucala R, Shimizu H. Topical application of anti-angiogenic peptides based on pigment epithelium-derived factor can improve psoriasis. J Dermatol Sci. 2010 Mar;57(3):183-91. doi: 10.1016/j.jdermsci.2009.12.010. Epub 2010 Jan 8. PMID 20060688
- [Result] Pyla R, Poulose N, Jun JY, Segar L. Expression of conventional and novel glucose transporters, GLUT1, -9, -10, and -12, in vascular smooth muscle cells. Am J Physiol Cell Physiol. 2013 Mar;304(6):C574-89. doi: 10.1152/ajpcell.00275.2012. Epub 2013 Jan 9. PMID 23302780
- [Result] Shurman DL, Glazewski L, Gumpert A, Zieske JD, Richard G. In vivo and in vitro expression of connexins in the human corneal epithelium. Invest Ophthalmol Vis Sci. 2005 Jun;46(6):1957-65. doi: 10.1167/iovs.04-1364. PMID 15914609
- [Derived] Mohany KM, Elkady S, Youssef EMK, Sayed NM, Idriss NK. Pigment epithelium-derived factor (PEDF) represses the glucose transporter 1 (GLUT1) mRNA expression and may be a potential therapeutic agent in psoriasis: a case-control and experimental study. Sci Rep. 2023 Dec 5;13(1):21424. doi: 10.1038/s41598-023-48565-9. PMID 38052851